CLINICAL TRIAL: NCT04942496
Title: A 96 Hour Patch Test Study Using Health Human Volunteers to Assess the Skin Irritation Potential of 11 Topically Applied Formulations
Brief Title: A 96-hour Patch Test Study Using Healthy Human Volunteers to Assess the Skin Irritation Potential of 11 Topically Applied Formulations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Molnlycke Health Care AB (Industry)
Collaborators: BioScience Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: #2011852-304
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Skin Irritancy Potential
MeSH Terms: interventions — chlorhexidine gluconate; long-chain-aldehyde dehydrogenase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (11):
- Test Product 1 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 2 (2% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 3 (2% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 4 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate; Device: Hibi Universal Bathing System
- Test Product 5 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 6 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 7 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 8 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- Test Product 9 (4% CHG) (Active Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back
  Interventions: Drug: Chlorhexidine Gluconate
- 0.1% Sodium Lauryl Sulfate (Placebo Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back. Product with known irritancy potential.
  Interventions: Other: 0.1% SLS
- Distilled Water (Placebo Comparator): Product applied to patch and randomly assigned application site on right and left parascapular regions of upper back. Product known not to cause irritancy
  Interventions: Other: Distilled Water

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Antimicrobial Skin Wash
  Arms: Test Product 1 (4% CHG); Test Product 2 (2% CHG); Test Product 3 (2% CHG); Test Product 4 (4% CHG); Test Product 5 (4% CHG); Test Product 6 (4% CHG); Test Product 7 (4% CHG); Test Product 8 (4% CHG); Test Product 9 (4% CHG)
Device: Hibi Universal Bathing System — Cloths used for patient bathing
  Arms: Test Product 4 (4% CHG)
Other: 0.1% SLS — Positive control
  Arms: 0.1% Sodium Lauryl Sulfate
Other: Distilled Water — Negative Control
  Arms: Distilled Water

SUMMARY:
This study is an evaluation of the irritation potential of 9 test products and 2 control materials applied to the backs of at least 44 volunteer human subjects over the course of a 96-hour period to determine and compare irritation scores. Subjects will be required to complete a 7-day pre-test conditioning period prior to the test period. Finn Chambers® on Scanpor® will be used to apply each test material to a designated site on the skin of the parascapular region of the upper back every 24 hours for 96 hours. The sites will be evaluated visually prior to the first patch application and immediately following each patch removal. Instrument measurements of transepidermal water loss (TEWL) will also be performed prior to the first patch application and will start between 15 to 30 minutes, following removal of each patch.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least at least 18 years of age but no more than 70 years of age, and of any race. Subjects that are 66 to 70 years of age are only eligible with proof of vaccination for COVID-19 having been completed at least 30 days prior to enrolling in the study.
* Subjects must be able to read and understand English.
* Subject's must have test sites on the skin of the back free of injury and in good condition (no active skin rashes, moderate to severe acne, tattoos on test areas, excessive hair, sunburn, excessive freckling, moles, scratches, breaks in the skin, etc.) and have no currently active skin diseases or skin conditions (for example, psoriasis, eczema) that may compromise subject safety or study integrity.
* Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, congenital heart disease, an organ transplant, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an immunocompromised condition such as AIDS (or HIV positive), lupus, fibromyalgia, ulcerative colitis, Crohn's disease, asthma, heart disease, hypertension, or medicated multiple sclerosis.
* Subjects must have read and signed the Informed Consent Form, List of Restricted Products, and Allowed and Restricted Products For Hand Cleaning During Coronavirus Disease 2019 (COVID-19) Pandemic prior to participating in the study, all located in the separate Informed Consent documents. Subjects must also have a current Authorization to Use and Disclose Protected Health Information Form on file at the testing facility.

Exclusion Criteria:

* Have participated in a clinical study in the past 7 days or be currently participating in another clinical study.
* Be experiencing any signs/symptoms of respiratory illness, including cough, fever (body temperature of ≥ 100.0 °F) or chills, shortness of breath or difficulty breathing, persistent pain or pressure in the chest, confusion or inability to respond to external stimuli, bluish lips/face, loss of taste/smell, sore throat, headache, nasal discharge ("runny nose"), frequent sneezing, or general fatigue / body aches.
* Have a current diagnosis of active Coronavirus Disease 2019 (COVID-19) or have been in close contact within the last 2 weeks of anyone who has been diagnosed as having contracted COVID-19.
* Have limited mobility that would hamper their ability to lay on their stomach for 45 minutes to an hour as directed.
* Have known allergies or sensitivities to latex (rubber), alcohols, sunscreens, deodorants, laundry detergents, topically applied fragrances, cleansers, soaps, lotions, or to common antibacterial agents, particularly chlorohexidine gluconate.
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin with the exception of plants known to cause reactions for most humans (e.g., poison oak or poison ivy).
* Have a known hypersensitivity to the test product or any of its components, especially in those with a history of possible chlorhexidine-related allergic reactions.
* Subjects must not be receiving any antihistamines, or anti-inflammatory medications in the 48 hours prior to testing through completion of the study.

Note - 81 mg of aspirin for preventative health reasons does not reduce inflammatory responses, and as such is not considered to be an exclusion to testing.

* Be receiving any antibiotic medications during the 7-day pre-test period through completion of the study.
* Be receiving any topical or systemic corticosteroids, steroids (including steroid medications used to treat asthma) other than for contraception, hormone therapy, or menopausal purposes during the 7-day pre-test period through completion of the study.
* Have any type of port (or portacath) or Peripherally Inserted Central Catheter (PICC).
* Be nursing a child.
* Be pregnant, plan to become pregnant or impregnate a sexual partner within the pre-test period through completion of the study.
* Have any medical condition or use any medications that, in the opinion of the Principal Investigator, or Consulting Physician(s) should preclude participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Visual Evaluation of Skin Condition | assessed every 24 hours for a total of 96 hours
  The grading scale for skin condition is from 0-7 (0 - no evidence of irritation and 7-a strong reaction spreading beyond the test site) Reapplication stopped for any grade above 3.

SECONDARY OUTCOMES:
Transepidermal water loss | assessed every 24 hours for a total of 96 hours
  By quantitating the rate of water evaporation of the skin using a multi probe adapter system and Tewameter (r) TM 300 probe

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Drake, Principal Investigator — BSLI
Locations (1):
- Bioscience Laboratories, Inc, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No